CLINICAL TRIAL: NCT01477619
Title: An Open-label, Single Dose, Parallel Group Study to Assess the Effects of Smoking Status, Age and Body Size on the Pharmacokinetics, Safety, and Tolerability of Tasimelteon in Healthy Volunteers
Brief Title: Effects of Smoking, Age and Body Size on Pharmacokinetics, Safety and Tolerability on Tasimelteon in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: VP-VEC-162-1107
Record Dates: First submitted 2011-11-17; First posted 2011-11-22 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics
MeSH Terms: interventions — tasimelteon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Smokers (Experimental): Split into BMI categories
  Interventions: Drug: Tasimelteon
- Non-Smokers (Experimental): Gender, age, and BMI matched to Smokers
  Interventions: Drug: Tasimelteon
- Elderly (Experimental)
  Interventions: Drug: Tasimelteon

INTERVENTIONS:
Drug: Tasimelteon — 20mg single dose on Day 1
  Other Names: VEC-162; BMS-214778

SUMMARY:
The purpose of this research study is to understand whether there is any difference in the amount of tasimelteon in the blood in smokers versus non-smokers. Additionally, this study will provide an assessment of the effect, if any, of age and body size on the safety and tolerability profile and the pharmacokinetics of tasimelteon.

ELIGIBILITY:
Inclusion Criteria:

Groups 1 and 2:

1. Men or women between 18 - 55 years, inclusive;
2. Smokers who test positive for cotinine at screening and baseline and smoke at least 10 cigarettes per day, for at least 6 months prior to screening (Group 1) OR Non-smokers [abstinence from smoking for at least 6 months before the screening visit and test negative for cotinine at screening and baseline (Group 2)] who are matched to Group 1 by gender, age (±10 years), and BMI category [underweight/normal (≤ 24.99), overweight (25.00-29.99), and obese (≥ 30.00)];
3. Males, non-fecund females (i.e., surgically sterilized, if procedure was done 6 months before screening or subject is postmenopausal, without menses for 6 months before screening), or females of child-bearing potential using an acceptable method of birth control for a period of 35 days before the first dosing and females must have a negative pregnancy test at the screening and baseline visits; Note 1: Acceptable methods of birth control include any one of the following: abstinence, vasectomized sexual partner, hormonal methods (i.e. pill, hormonal IUD, Depo-Provera, implants, patch, intravaginal device [NuvaRing]), intrauterine device (IUD [copper banded coils]), diaphragm, cervical cap, or condom with spermicidal jelly or foam.
4. Vital signs (after 3 minutes resting in a semi-supine position) which are within the ranges shown below:

   * Body temperature between 35.0-37.5 °C;
   * Systolic blood pressure between 90-150 mmHg;
   * Diastolic blood pressure between 50-95 mmHg;
   * Pulse rate between 50-100 bpm.

Group 3:

1. Men or women 65 years of age or older;
2. Non-smokers (abstinence from smoking for at least 6 months before the start of the study and test negative for cotinine at screening and baseline);
3. Vital signs (after 3 minutes resting in a semi-supine position) which are within the ranges shown below:

   * Systolic blood pressure between 90-160 mmHg;
   * Diastolic blood pressure between 50-99 mmHg;
   * Pulse rate between 50-100 bpm.

Groups 1-3:

1. Ability and acceptance to provide written informed consent;
2. Willing and able to comply with study requirements and restrictions;
3. Subjects must be in good health as determined by past medical history, physical examination, electrocardiogram, clinical laboratory tests and urinalysis;

Exclusion Criteria:

1. History of recent (within six months) drug or alcohol abuse as defined in DSM IV, Diagnostic Criteria for Drug and Alcohol Abuse or evidence of such abuse as indicated by the laboratory assays conducted during the Screening Visit or at Baseline;
2. Any major surgery within three months of Baseline or any minor surgery within one month;
3. History or current evidence of cardiovascular, hepatic, hematopoietic, renal, gastrointestinal or metabolic dysfunction judged by the Investigator to be clinically significant;
4. Any condition requiring the regular use of medication except those listed in Section 8.2;
5. Use of any melatonin preparation chronically within 2 months prior to Day 1 or any drug known to cause major organ system toxicity (e.g., chloramphenicol or tamoxifen) within 60 days prior to Day 1.
6. Exposure to any investigational drug, including placebo, within 30 days or 5 half-lives (whichever is longer) of baseline;
7. Donation or loss of 400 mL or more of blood within two months prior to the Baseline Visit;
8. Significant illness within the two weeks prior to Baseline;
9. A known hypersensitivity to tasimelteon or drugs similar to tasimelteon including melatonin;
10. Pregnant or lactating females;
11. History of liver disease and/or positive for one or more of the following serological results:

    * A positive hepatitis C antibody test (anti-HCV)
    * A positive hepatitis B surface antigen (HBsAg)
12. A positive HIV test result
13. Any surgical or medical condition which might significantly alter the absorption, distribution or excretion of any drug. The Investigator should be guided by evidence of any of the following:

    * Clinically significant gastritis, ulcers, gastrointestinal or rectal bleeding within 5 years of the screening visit;
    * History of inflammatory bowel syndrome, major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection;
    * Pancreatic injury or pancreatitis within 5 years of the screening visit;
    * Clinically significant urinary obstruction or difficulty voiding within 3 years of the screening visit;
14. Exposure (within 2 weeks of the Baseline Visit) of any over-the-counter medications including dietary supplements and/or herbal remedies, except those listed in Section 8.2;
15. Use of any food or beverage containing grapefruit or grapefruit juice, apple or orange juice, vegetables from the mustard green family (e.g. kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard greens) and charbroiled meats for at least 2 weeks before the Baseline Visit until the end of the study;
16. Inability to be venipunctured and/or tolerate venous access;
17. Subjects who are unable to read or speak English;
18. Participation in a previous BMS-214778/VEC-162 trial;
19. Any other sound medical reason as determined by the clinical Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Tasimelteon plasma concentrations and pharmacokinetics in smokers versus non-smokers | Day 1 - Day 2
  Plasma concentrations and pharmacokinetics of tasimelteon of group 1 (smokers) will be compared to group 2 (non-smokers)
To assess the effect of weight, body mass index (BMI), and age on the pharmacokinetic profile of tasimelteon | Day 1 -Day 2
  Pharmacokinetics of tasimelteon will be compared using all three groups (smokers, non-smokers and elderly). Group 1 and Group 2 will be gender, age and BMI category matched.

SECONDARY OUTCOMES:
To assess plasma concentrations and pharmacokinetics of tasimelteon metabolites (M3, M9, M11, M12, M13, and M14) in subjects who smoke compared to subjects who do not smoke. | Day 1 - Day 2
  Composite of 24 hour pharmacokinetic parameters will be compared between group 1 (smokers) and group 2 (non-smokers)
To assess the effect of weight, BMI, and age on the pharmacokinetic profile of tasimelteon metabolites (M3, M9, M11, M12, M13, and M14). | Day 1 - Day 2
  Composite of 24 hour pharmacokinetic parameters will be compared using all three groups (smokers, non-smokers and elderly). Group 1 and Group 2 will be gender, age and BMI category matched.
Tasimelteon safety and tolerability | Day 1
  Safety of single dose as measured by adverse event reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Vanda Pharmaceuticals, Study Director — Vanda Pharmaceuticals
Locations (1):
- Bio-Kinetic Clinical Applications, Springfield, Missouri, United States